CLINICAL TRIAL: NCT07140744
Title: A Prospective Diagnostic Study Evaluating the Impact of P-tau217 Blood Biomarker Testing on Early Evaluation and Management of Patients Presenting With Cognitive Complaint in Primary and Secondary/Tertiary Care
Brief Title: A Study Evaluating the Impact of P-tau217 Blood Biomarker Testing on Early Evaluation and Management of Patients Presenting With Cognitive Complaint
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 28782; J4Y-MC-S003 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Subjective Cognitive Impairment
Keywords: Diagnostic utility; Blood biomarkers; Blood diagnostics
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Other): Stratified by Primary Care Physician (PCP) versus Secondary/Tertiary Physician (S/TCP)
  Patient participants in the interventional group will undergo P-tau217 testing.
  Interventions: Diagnostic Test: P-tau217
- Standard of Care Group (Other): Stratified by PCP versus S/TCP
  Patient participants in the standard of care group (SOC) will not undergo sponsor-provided P-tau217 testing.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Diagnostic Test: P-tau217 — Blood biomarker testing
  Arms: Interventional Group
Other: Standard of Care — Standard of care
  Arms: Standard of Care Group

SUMMARY:
The purpose of the study is to measure the difference in the proportion of participants with prespecified patient management actions between a tested interventional group and a control group.

DETAILED DESCRIPTION:
There are two types of participants in this study, HCP participants and patient participants. Outcome measures relate to the HCP management of patient participants.

ELIGIBILITY:
Inclusion Criteria:

Health Care Provider (HCP) Definitions

* Primary care physician (PCPs): physicians such as family medicine practitioners and internists who do not specialize in neurological care.
* Secondary care physicians (SCPs): physicians such as geriatricians or neurologists who see patients for specific reasons.
* Tertiary care physicians (TCPs): specialty neurologists who focus on certain neurological conditions.

HCP Participant Selection Criteria

* HCP inclusion criterion for each category of HCP is as follows:

  * Group 1: PCPs who routinely evaluate and manage patients over the age of 50 in a family practice or internist setting.
  * Group 2: SCPs and TCPs with experience diagnosing and treating patients with cognitive impairment and dementia.

Additional inclusion criteria applying to HCPs in the interventional group:

* Must be willing to review educational materials provided by the study sponsor, before enrolling patients.

Patient Participant Criteria

* Participants in the interventional group are eligible to be included in the study only if all the following criteria apply:

  * Are capable of giving, and have given, signed informed consent.
  * Have venous access sufficient to allow the protocol-required blood sampling.
  * Are reliable, willing, and able to make themselves available for the duration of the study and are willing to follow study procedures.

Disease-specific Characteristics

* Present to the HCP with 1 or more subjective cognitive impairment complaints (SCIC) in the 4 weeks prior to identification: for example, worsening of memory, misplacing items, difficulty concentrating, or new challenges with problem solving.

Patient Participant Exclusion Criteria:

* In the 18 months prior to identification have prior or associated HCP-ordered referral or prior prescription of drug therapies, for the SCIC
* Participants with previous amyloid- or tau-specific tests, defined as

  * Amyloid position emission tomography (PET)
  * Tau PET
  * Cerebral spinal fluid (CSF) tests for amyloid beta (Aβ) and/or tau biomarkers, or
  * Blood tests for Aβ and/or tau biomarkers
* Has a current serious or unstable illness that in the enrolling investigator's opinion could interfere with completion of the study or have a life expectancy of less than 1 year.
* Has a known brain lesion, pathology, or prior alternative diagnosis that could explain the participant's clinical presentation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Difference in Proportion of Participants Between the Primary Care Physician (PCP) Tested Group and the PCP Control Group with at Least 1 Management Action | 6 Months
  Difference in proportion of participants with a least 1 management action, referral to Secondary or Tertiary Care Physician (S/TCP); counseling; Alzheimer's Disease (AD) drug therapy related to cognitive complaint, or Non-AD drug therapy related to cognitive complaint.

SECONDARY OUTCOMES:
Difference in Proportion of Participants Between the S/TCP Tested Group and the S/TCP Control Group with at Least 1 Management Action | 6 and 12 Months
  Difference in proportion of participants with a least 1 management action, referral to S/TCP; counseling; AD drug therapy related to cognitive complaint, or Non-AD drug therapy related to cognitive complaint.
Time from Cognitive Complaint to Date of Referral to a S/TCP Between the PCP Tested Group and the PCP Control Group: | 6 and 12 Months
Time from Cognitive Complaint to Date of Counseling Between the PCP Tested Group and the PCP Control Group | 6 and 12 Months
Time from Cognitive Complaint to Date of Initiating AD Therapy Between the PCP Tested Group and the PCP Control Group | 6 and 12 Months
Time from Cognitive Complaint to Date of Initiating Non-AD Therapy Between the PCP Tested Group and the PCP Control Group | 6 and 12 Months
Time from Cognitive Complaint to Date of Referral to a S/TCP Between the S/TCP Tested Group and the S/TCP Control Group: | 6 and 12 Months
Time from Cognitive Complaint to Date of Counseling Between the S/TCP Tested Group and the S/TCP Control Group | 6 and 12 Months
Time from Cognitive Complaint to Date of Initiating AD Therapy Between the S/TCP Tested Group and the S/TCP Control Group | 6 and 12 Months
Time from Cognitive Complaint to Date of Initiating Non-AD Therapy Between the S/TCP Tested Group and the S/TCP Control Group | 6 and 12 Months
Difference in Proportion of Participants with a Documented Alzheimer's Disease-Specific International Classification of Diseases (ICD) - 10 Code Between the S/TCP Tested Group and the S/TCP Control Group | 6 and 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- SiteRx Virtual Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/